CLINICAL TRIAL: NCT02433678
Title: An Investigation Into The Anti-hypertensive And Potential Anti-inflammatory Actions Of Dapagliflozin
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University at Buffalo (Other)
Collaborators: Kaleida Health (Other)
Responsible Party: Principal Investigator, Paresh Dandona, distinguished professor, University at Buffalo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1972
Record Dates: First submitted 2015-04-24; First posted 2015-05-05 (Estimated); Results first posted 2019-10-30 (Actual); Last update posted 2019-10-30 (Actual); Status verified 2019-10

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — dapagliflozin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Patients will be treated for 12 weeks with placebo once daily
  Interventions: Drug: Placebo
- Dapagliflozin (Active Comparator): 10 mg daily for the 12 weeks
  Interventions: Drug: dapagliflozin

INTERVENTIONS:
Drug: dapagliflozin — SGLT-2 inhibitor for the treatment of type 2 diabetes
  Other Names: Farxiga
  Arms: Dapagliflozin
Drug: Placebo
  Arms: Placebo

SUMMARY:
This is a single center, prospective, randomized, placebo -controlled, parallel design and double blind study to evaluate oxidative stress, inflammation and hypertension markers and mediators before and after treatment with dapagliflozin.

DETAILED DESCRIPTION:
Two groups of 26 patients each (total 52 patients) with type 2 diabetes on oral agents will be included in the study. One group will be randomized to dapagliflozin (a dose of 5 mg daily will be titrated to 10 mg daily during the first week) while the other will be placebo. The patients will be treated for 12 weeks. Only half the patients (equal numbers in both groups) will be tested for the secondary endpoints related to postprandial and single dose induced changes. The primary endpoint of the study is to detect a significant difference in the percent change in fasting Nuclear factor-k B (NFκB) activation (DNA binding activity) in mononuclear cells (MNC) before and after dapagliflozin use (0 week vs. 12 weeks) as compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

* Age 20-80 years inclusive.
* Type 2 diabetes
* BMI ≥30 kg/m2
* Subjects on statins, ACE inhibitors, ARBs, thiazolidinediones and -antioxidants will be allowed as long as they are on stable doses of these -compounds and the dosage in not changed during the course of study. -Patients will be evenly distributed between the 2 groups based on statins, -ARBs, TZDs and ACE inhibitors use.
* HbA1c ≤ 8.0%

Exclusion Criteria:

* Use of GLP-1 agonists or DPP-IV or SGLT-2 inhibitors therapy in the last 3 -months.
* Risk for pancreatitis, i.e., history of gallstones, alcohol abuse, and -hypertriglyceridemia.
* Coronary event or procedure (myocardial infarction, unstable angina, coronary -artery bypass, surgery or coronary angioplasty) in the previous 3 months.
* Hepatic disease: Severe hepatic insufficiency and/or significant abnormal liver -function defined as:
* aspartate aminotransferase (AST) >3x upper limit of normal (ULN) and/or -alanine aminotransferase (ALT) >3x ULN
* Total bilirubin >2.0 mg/dL (34.2 µmol/L)
* Positive serologic evidence of current infectious liver disease including Hepatitis B viral antibody IGM, Hepatitis B surface antigen and Hepatitis C virus antibody
* (liver function tests more than 3 times the upper limit of normal)
* Renal impairment (serum eGFR <60 ml/min)
* Any other life-threatening, non-cardiac disease
* Uncontrolled hypertension (BP > 160/100 mm of Hg)
* Congestive Heart Failure class III or IV.
* Use of an investigational agent or therapeutic regimen within 30 days of study
* Participation in any other concurrent clinical trial
* pregnant or breastfeeding patients
* Volume depleted patients. Patients at risk for volume depletion due to co-existing conditions or concomitant medications, such as loop diuretics

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2015-11; Primary Completion 2018-03 (Actual); Study Completion 2018-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paresh Dandona, MD, PhD, Principal Investigator — University at Buffalo
Locations (1):
- ECMC Ambulatory Center, 3rd Floor, Buffalo, New York, United States

REFERENCES:
- [Derived] Ghanim H, Abuaysheh S, Hejna J, Green K, Batra M, Makdissi A, Chaudhuri A, Dandona P. Dapagliflozin Suppresses Hepcidin And Increases Erythropoiesis. J Clin Endocrinol Metab. 2020 Apr 1;105(4):dgaa057. doi: 10.1210/clinem/dgaa057. PMID 32044999

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Patients will be treated for 12 weeks with placebo once daily
  Placebo
Period: Overall Study
Arm/Group | Placebo | Dapagliflozin
Started | 26 | 26
Completed | 25 | 24
Not Completed | 1 | 2
Not completed — Lost to Follow-up | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Dapagliflozin | Total
Number analyzed (Participants) | 26 | 26 | 52
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 16 | 22 | 38
  >=65 years | 10 | 4 | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 61 (10) | 61 (9) | 61 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 11 | 19
  Male | 18 | 15 | 33
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 8 | 8 | 16
  White | 18 | 17 | 35
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 26 | 26 | 52

OUTCOME MEASURES:

1. Primary Outcome: Difference in the Percent Change in Fasting Nuclear Factor Kappa-light-chain-enhancer of Activated B Cells Activation (DNA Binding Activity) in Mononuclear Cells Before and After Dapagliflozin Use
Description: nuclear factor kappa-light-chain-enhancer of activated B cells measurement through Transcription factor assay
Time Frame: 12 weeks
Population: Out of the 26 total patients in each group, 4 dropped in the placebo arm and 3 dropped in the Dapagliflozin arm
Measure: Mean (Standard Deviation); unit: arbitrary unit
Arm/Group | Placebo | Dapagliflozin
Number analyzed (Participants) | 22 | 23
arbitrary unit
  baseline | 0.762 (0.14) | 0.733 (0.11)
  6 week | 0.802 (0.12) | 0.835 (0.13)
  12 week | 0.776 (0.15) | 0.815 (0.12)

2. Secondary Outcome: Changes in Expression of Inflammatory Mediators
Description: p47phox in mononuclear cells through real time polymerase chain reaction
Time Frame: 12 Weeks
Population: Out of the 26 total patients in each group, 4 dropped in the placebo arm and 3 dropped in the Dapagliflozin arm
Measure: Mean (Standard Deviation); unit: arbitrary unit
Arm/Group | Placebo | Dapagliflozin
Number analyzed (Participants) | 22 | 23
arbitrary unit
  baseline | 100 (0) | 100 (0)
  12 week | 92 (14) | 104 (12)

3. Secondary Outcome: Changes in Expression of Inflammatory Mediators
Description: Suppressor Of Cytokine Signaling 3 measurement in Mononuclear cells through real time polymerase chain reaction
Time Frame: 12 weeks
Population: Out of the 26 patients in each group, 4 dropped in the placebo arm and 3 dropped in the drug arm
Measure: Mean (Standard Deviation); unit: arbitrary unit
Arm/Group | Placebo | Dapagliflozin
Number analyzed (Participants) | 22 | 23
arbitrary unit
  baseline | 0.72 (0.20) | 0.60 (0.17)
  12 week | 0.70 (0.19) | 0.66 (0.19)

4. Secondary Outcome: Changes in Expression of Inflammatory Mediators
Description: Interleukin 1 Beta measurement in mononuclear cells through real time polymerase chain reaction
Time Frame: 12 weeks
Population: Out of the 26 patients in each group, 4 dropped in the placebo arm and 3 dropped in the drug arm
Measure: Mean (Standard Deviation); unit: arbitrary unit
Arm/Group | Placebo | Dapagliflozin
Number analyzed (Participants) | 22 | 23
arbitrary unit
  baseline | 0.697 (0.21) | 0.756 (0.19)
  12 week | 0.705 (0.21) | 0.741 (0.17)

5. Secondary Outcome: Changes in Expression of Inflammatory Mediators
Description: c-Jun N-terminal kinase 1 measurement in Mononuclear cells through real time polymerase chain reaction
Time Frame: 12 weeks
Population: Out of the 26 patients in each group, 4 dropped in the placebo arm and 3 dropped in the drug arm
Measure: Mean (Standard Deviation); unit: arbitrary unit
Arm/Group | Placebo | Dapagliflozin
Number analyzed (Participants) | 22 | 23
arbitrary unit
  baseline | 0.802 (0.19) | 0.856 (0.20)
  12 week | 0.810 (0.21) | 0.820 (0.19)

6. Secondary Outcome: Changes in Expression of Inflammatory Mediators
Description: Toll-like receptor 4 measurement in mononuclear cells through real time polymerase chain reaction
Time Frame: 12 weeks
Population: Out of the 26 patients in each group, 4 dropped in the placebo arm and 3 dropped in the drug arm
Measure: Mean (Standard Deviation); unit: arbitrary unit
Arm/Group | Placebo | Dapagliflozin
Number analyzed (Participants) | 22 | 23
arbitrary unit
  baseline | 0.704 (0.15) | 0.774 (0.21)
  12 week | 0.708 (0.17) | 0.731 (0.13)

7. Secondary Outcome: Changes in Expression of Inflammatory Mediators
Description: Tumor necrosis factor alpha measurement in mononuclear through real time polymerase chain reaction
Time Frame: 12 weeks
Population: Out of the 26 patients in each group, 4 dropped in the placebo arm and 3 dropped in the drug arm
Measure: Mean (Standard Deviation); unit: arbitrary unit
Arm/Group | Placebo | Dapagliflozin
Number analyzed (Participants) | 22 | 23
arbitrary unit
  baseline | 0.762 (0.14) | 0.733 (0.11)
  12 week | 0.776 (0.15) | 0.815 (0.12)

8. Other Pre Specified Outcome: Change in Hypertension Mediators
Description: Plasma concentrations measurement of Angiotensinogen through enzyme-linked immunosorbent assay
Time Frame: 12 weeks
Population: Out of the 26 patients in each group, 4 dropped in the placebo arm and 3 dropped in the drug arm
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | Placebo | Dapagliflozin
Number analyzed (Participants) | 22 | 23
ug/mL
  baseline | 7.08 (0.41) | 7.23 (0.60)
  12 week | 6.98 (0.38) | 5.88 (0.64)

9. Other Pre Specified Outcome: Change in Hypertension Mediators
Description: Plasma concentration measurement of Angitosensin II through enzyme-linked immunosorbent assay
Time Frame: 12 weeks
Population: Out of the 26 patients in each group, 4 dropped in the placebo arm and 3 dropped in the drug arm
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Placebo | Dapagliflozin
Number analyzed (Participants) | 22 | 23
pg/mL
  baseline | 24.5 (5.5) | 29.2 (6.5)
  12 week | 25.1 (5.9) | 19.6 (7.0)

10. Other Pre Specified Outcome: Change in Hypertension Mediators
Description: Plasma concentration measurement of Renin through enzyme-linked immunosorbent assay
Time Frame: 12 weeks
Population: Out of the 26 patients in each group, 4 dropped in the placebo arm and 3 dropped in the drug arm
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Placebo | Dapagliflozin
Number analyzed (Participants) | 22 | 23
pg/mL
  baseline | 1599 (492) | 1630 (133)
  12 week | 1632 (543) | 1844 (145)

11. Other Pre Specified Outcome: Change in Hypertension Mediators
Description: Plasma concentration measurement of Atrial natriuretic peptide through enzyme linked immunosorbent assay
Time Frame: 12 weeks
Population: Out of the 26 patients in each group, 4 dropped in the placebo arm and 3 dropped in the drug arm
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Placebo | Dapagliflozin
Number analyzed (Participants) | 22 | 23
pg/mL
  baseline | 83 (12) | 92 (8)
  12 week | 86 (18) | 125 (37)

12. Other Pre Specified Outcome: Change in Hypertension Mediators
Description: Plasma concentration measurement of B-type natriuretic peptide through enzyme linked immunosorbent assay
Time Frame: 12 weeks
Population: Out of the 26 patients in each group, 4 dropped in the placebo arm and 3 dropped in the drug arm
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Placebo | Dapagliflozin
Number analyzed (Participants) | 22 | 23
pg/mL
  baseline | 59.2 (12.9) | 64.7 (13.7)
  12 week | 64.3 (20.1) | 62.9 (13.8)

13. Other Pre Specified Outcome: Change in Hypertension Mediators
Description: Plasma concentration measurement of Cyclic guanosine monophosphate through enzyme linked immunosorbent assay
Time Frame: 12 weeks
Population: Out of the 26 patients in each group, 4 dropped in the placebo arm and 3 dropped in the drug arm
Measure: Mean (Standard Deviation); unit: pmol/mL
Arm/Group | Placebo | Dapagliflozin
Number analyzed (Participants) | 22 | 23
pmol/mL
  baseline | 64 (18) | 73 (11)
  12 week | 73 (22) | 89 (12)

14. Other Pre Specified Outcome: Change in Hypertension Mediators
Description: Plasma concentration measurment of Cyclic adenosine monophosphate through enzyme linked immunosorbent assay
Time Frame: 12 week
Population: Out of the 26 patients in each group, 4 dropped in the placebo arm and 3 dropped in the drug arm
Measure: Mean (Standard Deviation); unit: pmol/mL
Arm/Group | Placebo | Dapagliflozin
Number analyzed (Participants) | 22 | 23
pmol/mL
  baseline | 80 (4) | 78 (5)
  12 week | 77 (5) | 80 (5)

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Placebo | Dapagliflozin
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/26
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/26
Other Adverse Events (participants affected / at risk) | 0/26 | 0/26

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2018-10-02): https://cdn.clinicaltrials.gov/large-docs/78/NCT02433678/Prot_000.pdf